CLINICAL TRIAL: NCT03520868
Title: Heparin Requirements in Patients Undergoing Atrial Fibrillation Ablation on Coumadin vs NOACs
Status: Completed | Type: Observational
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Responsible Party: Principal Investigator, Michael Orlov, Electrophysiologist, Steward St. Elizabeth's Medical Center of Boston, Inc.
Other Study IDs: 00747
Record Dates: First submitted 2017-10-31; First posted 2018-05-11 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum blood test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Coumadin: Coumadin patients with undergo standard procedure with monitoring of Anti-Factor Xa assay level before and during the procedure. Heparin bolus given will be based on 70 U/kg
  Interventions: Diagnostic Test: Monitoring Anti Factor Xa level
- Dabigatran: Dabigatran patients with undergo standard procedure with monitoring of Anti-Factor Xa assay level before and during the procedure. Heparin bolus given will be based on 110 U/kg
  Interventions: Diagnostic Test: Monitoring Anti Factor Xa level
- Rivaroxiban: Rivaroxiban patients with undergo standard procedure with monitoring of Anti-Factor Xa assay level before and during the procedure. Heparin bolus given will be based on 110 U/kg
  Interventions: Diagnostic Test: Monitoring Anti Factor Xa level
- Apixaban: Apixaban patients with undergo standard procedure with monitoring of Anti-Factor Xa assay level before and during the procedure. Heparin bolus given will be based on 10 U/kg
  Interventions: Diagnostic Test: Monitoring Anti Factor Xa level

INTERVENTIONS:
Diagnostic Test: Monitoring Anti Factor Xa level — Each patient will have baseline Anti-Factor Xa assay checked. During the procedure, Anti-Factor Xa assay is checked concurrently with ACT after heparin bolus and infusion.

SUMMARY:
To observe, using a prospectively designed study, the effect of type of oral anticoagulant on intra-procedural heparin requirements in patients undergoing Atrial Fibrillation ablation and to assess whether ACT assay accurately reflects heparin anti coagulation effect.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia affecting the US population and accounts for 15% of strokes worldwide. Radiofrequency ablation has become a frequently used therapy for treatment of afib after failure of at least one anti-arrhythmic drug. Pulmonary Vein Isolation (PVI) remains the cornerstone of AF ablation and requires transseptal puncture and placement of catheters in the left atrium which can be thrombogenic and cause stroke. This is avoided by intra-procedural infusion of heparin and the anti-coagulation effect is monitored using Activated Clotting Time (ACT). With the approval of Novel Oral Anti-Coagulants (NOAC), increasing number of patients are undergoing AF ablation on these medications. It has been observed that patients on NOACs require much larger doses of heparin and take longer time to reach therapeutic ACT. Consequently, patients are at higher risk for thromboembolism and stroke. On the other hand, higher doses of heparin can expose patients to excessive bleeding complications. The investigators seek to explain the mechanism of "heparin resistance" in such a patient population and to develop a protocol that can achieve therapeutic anticoagulation quicker.

ELIGIBILITY:
Inclusion Criteria:

* All adults, male and female, aged 18 and above.
* Patients with paroxysmal, persistent or chronic AF
* All patients must be on therapeutic doses of Coumadin or one of the NOACs for at least 1 month prior to the procedure.

Exclusion Criteria:

* Patients with known primary or secondary coagulopathy (such as Hemophilia, vWF deficiency, active malignancy, ATIII deficiency, Factor V Leiden deficiency, Hx of recurrent DVT/PE)
* Patients with hypoalbuminemia, cirrhosis
* chronic LMWH therapy,
* ESRD on HD, and severely impaired kidney function with CKD stage IV
* BMI >35
* prosthetic heart valves and
* advanced liver disease
* previous procedural complications such as tamponade

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults, male and female, aged 18 and above, who have been referred to the EP lab for elective PVI (Pulmonary Vein Isolation).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Intra-procedural Heparin Requirements in patients taking NOACs and Coumadin | During the procedure
  The investigators will measure the amount of intravenous heparin administered to each patient during the afib ablation to achieve therapeutic anticoagulation.

SECONDARY OUTCOMES:
Anti Factor Xa assay measured to assess Heparin activity during Atrial Fibrillation Ablation | During the procedure
  The intra-procedural heparin activity is measured using Anti Factor Xa assay.
Activated Clotting Time (ACT) measured to assess Heparin activity during Atrial Fibrillation Ablation | During the procedure
  The intra-procedural heparin activity is measured using ACT

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Orlov, MD, Principal Investigator — Steward St. Elizabeth's Medical Center of Boston, Inc.
Locations (1):
- St Elizabeth Medical Center, Brighton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No